CLINICAL TRIAL: NCT04596826
Title: The Effect of Dronabinol on Ocular Hemodynamics in Patients With Primary
Brief Title: The Effect of Dronabinol on Ocular Hemodynamics in Patients With Primary Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc. Prof. PD Doreen Schmidl, MD, PhD,, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: OPHT-250719
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-12

CONDITIONS: Retinal Blood Flow
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- healthy subjects (Experimental)
  Interventions: Drug: Dronabinol 5 MG; Drug: Dronabinol 10 MG; Drug: Placebo
- glaucoma patients (Experimental)
  Interventions: Drug: Dronabinol 5 MG; Drug: Dronabinol 10 MG; Drug: Placebo
- healthy volunteers (Placebo Comparator)
  Interventions: Drug: Dronabinol 5 MG; Drug: Dronabinol 10 MG; Drug: Placebo
- Glaucoma patients (Placebo Comparator)
  Interventions: Drug: Dronabinol 5 MG; Drug: Dronabinol 10 MG; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 5 MG — oral administration
Drug: Dronabinol 10 MG — oral administration
Drug: Placebo — oral administration

SUMMARY:
Glaucoma is among the leading causes for irreversible blindness worldwide. While lowering intraocular pressure (IOP) remains the mainstay of therapy, there are still some patients who progress despite well-controlled IOP. There is evidence from several studies that ocular blood flow and its regulation is impaired in patients with glaucoma. Tetrahydrocannabinol (THC) has been used in the treatment for glaucoma in some countries for several years due to its IOP lowering effect. In addition, there is also evidence that THC features neuroprotective effects and improves ocular hemodynamics. Dronabinol is a synthetic THC that is legally available in several European countries. It has the advantage that exact dosing of THC is possible in contrast to previously applied administration forms such as smoking. Due to its legal status in the past, data about the effect of THC on ocular blood flow and its regulation are sparse. In a recent study conducted in the investigators laboratory they found that single administration of dronabinol leads to a significant increase in optic nerve head (ONH) blood flow without impairing its autoregulatory capacity.The aim of the present study therefore is to investigate whether single administration of dronabinol alters optic nerve head (ONH) blood flow in patients with open angle glaucoma. In addition, other parameters for ocular blood flow will be measured, in particular retinal blood flow, retinal oxygen saturation and retinal neurovascular coupling. The study will be conducted in a parallel-group, randomized, double-masked, placebo-controlled, cross-over design. Patients will be randomized to either receive 5mg or 10mg dronabinol on one study day. Other studies investigating retinal hemodynamics or IOP after administration of THC also have used similar or slightly higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of manifest open angle glaucoma as defined as pathological optic disc appearance, glaucoma hemifield test outside normal limits and/or untreated IOP ≥ 21 mmHg on at least three measurements in the medical history.

  * Mean deviation in the visual field test < 10dB
  * Informed consent signed and dated
  * Patient aged ≥ 18 years old
  * Ametropia ≤ 6 diopters
  * Normal findings in the medical history and physical examination including ECG unless the investigator considers an abnormality to be clinically irrelevant
  * Normal findings in the laboratory testing unless the investigator considers an abnormality to be clinically irrelevant
  * Nonsmokers

Exclusion Criteria:

* Exfoliation glaucoma

  * Pigmentary glaucoma
  * Secondary glaucoma
  * History of acute angle closure
  * Intraocular surgery within the last 6 months
  * Filtration surgery for glaucoma at any time
  * Laser procedure for glaucoma within the last 12 months Visual field not performed or not available within 6 months
  * Ocular inflammation or infection within the last 3 months
  * Regular use of medication that potentially could interact with THC, abuse of alcoholic beverages or drugs
  * History of drug or alcohol abuse
  * Psychiatric disorders in the medical history
  * Risk for drug dependence as evaluated by a psychiatrist
  * Participation in a clinical trial in the 3 weeks preceding the study
  * Positive urine drug test at the screening examination or on the study days
  * Positive alcohol breath test at the screening examination or on the study days
  * Regular consumption of cannabis and inability to not consume cannabis during the study period
  * Symptoms of a clinically relevant illness in the 3 weeks before the first study day
  * History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
  * Blood donation during the previous 3 weeks
  * Known hypersensitivity to any of the components of the IMP under investigation or other study medication
  * History or family history of epilepsy
  * Pregnant or breast-feeding women
  * Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (oral contraceptives, intra-uterine device, contraceptive implant or condoms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow | 60 minutes on the study day
  To determine the total blood flow in the eye, OCT measurements were performed with a rectangular scanning pattern around the optical nerve head.

OTHER OUTCOMES:
Flicker induced increase in retinal blood flow using a Fourier Domain Doppler OCT | 30 minutes on the study day
Retinal vessel diameter (DVA) | 30 minutes on the study day
  The DVA allows for the real time measurement of retinal vessel diameters in vivo.
  The DVA is a commercially available system (IMEDOS, Jena, Germany) which comprises a fundus camera, a video camera, a real time monitor and a personal computer with an analyzing software for the accurate determination of retinal arterial and venous diameters. Every second a maximum of 25 readings of vessel diameter can be obtained. For this purpose the fundus is imaged onto the charge coupled device chip of the video camera. The consecutive fundus images are digitized using a frame grabber. In addition, the fundus image can be inspected on the real time monitor and, if necessary, stored on a video recorder. Evaluation of the retinal vessel diameters can either be done online or offline from the recorded video tapes
Retinal oxygen saturation (DVA) | 30 minutes on the study day
  In particular, retinal oxygen saturation measurement is based on the image analysis by the DVA software of two monochromatic fundus images as recorded by a standard DVA. In an image, obtained by the camera and filter assembly, the operator has to mark the vessel of interest by a mouse click. The vessel is traced automatically applying the following procedure. The vessel walls are located as photometric edges in the vicinity of the mouse cursor in the green channel image. If edges are determined, the search is continued in their proximity.
Retinal blood velocities | 15 minutes on the study day
  We observe bi-directional blood flow and pulsatility of blood velocity in retinal vessels with a Doppler detection bandwidth of 12.5 kHz and a longitudinal velocity sensitivity in tissue of 200μm/s.
THC plasma concentration | 120 minutes on the study day
  Measurements of ocular hemodynamics will be started one hour after administration, since maximum plasma levels are reached 60-120 minutes after administration.
Retinal vessel density (OCTA) | 30 minutes on the study day
Normalized blur (LSFG) | 15 minutes on the study day
Relative flow volume (LSFG) | 30 minutes on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Lindner T, Pai V, Janku P, Hommer N, Hommer A, Abensperg-Traun M, Petric L, Schmetterer L, Garhofer G, Schmidl D. Single oral administration of dronabinol increases ocular blood flow in patients with glaucoma. Acta Ophthalmol. 2026 Mar;104(2):225-232. doi: 10.1111/aos.17573. Epub 2025 Aug 7. PMID 40772417